CLINICAL TRIAL: NCT03255083
Title: A Multicenter, Open-Label Phase 1 Study of DS-1205c in Combination With Osimertinib in Subjects With Metastatic or Unresectable EGFR-Mutant Non-Small Cell Lung Cancer
Brief Title: DS-1205c With Osimertinib for Metastatic or Unresectable Epidermal Growth Factor Receptor (EGFR)-Mutant Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated based on a business decision by the Sponsor.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1205-A-U101
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Oncology; Advanced Non-small Cell Lung Cancer; Inoperable Non-small Cell Lung Cancer; Metastatic; Non-resectable; Epidermal growth factor receptor; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DS-1205c with osimertinib (Experimental): Participants receive DS-1205c (at planned doses given orally twice daily: 200 mg, 400 mg, 800 mg, 1200 mg) in combination with daily 80 mg oral dose of osimertinib
  Interventions: Drug: DS-1205c; Drug: Osimertinib

INTERVENTIONS:
Drug: DS-1205c — DS-1205c 200 mg capsule
Drug: Osimertinib — Osimertinib 80 mg tablet

SUMMARY:
This study has two parts: dose escalation and dose expansion.

The primary objectives are:

* For Dose Escalation, to assess the safety and tolerability of DS-1205c when combined with osimertinib in the study population and to determine the recommended dose for expansion of DS-1205c when combined with osimertinib in the study population
* For Dose Expansion, to assess the safety and tolerability of DS-1205c when combined with osimertinib in the study population

In Dose Escalation, after a 7-day run in period (Cycle 0), there will be 21-day cycles (Cycle 1 onward). In Dose Expansion, there will be 21-day cycles.

The number of treatment cycles is not fixed in this study. Participants will continue study treatment until they decide not to (withdraw consent), their disease gets worse [progressive disease (PD)], or side effects become unacceptable (unacceptable toxicity).

ELIGIBILITY:
Inclusion Criteria:

1. Has histologically or cytologically documented adenocarcinoma NSCLC.
2. Has locally advanced or metastatic NSCLC, not amenable to curative surgery or radiation.
3. Has acquired resistance to EGFR TKI according to the Jackman criteria (PMID: 19949011):

   1. Historical confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) or
   2. Has experienced clinical benefit from an EGFR TKI, followed by systemic progression (Response Evaluation Criteria in Solid Tumors [RECIST version 1.1] or World Health Organization [WHO]) while on continuous treatment with an EGFR TKI.
4. Is currently receiving, and is able to discontinue erlotinib, gefinitib, or afatinib; or is currently receiving osimertinib at the prescribed 80 mg dose and is able to interrupt osimertinib.
5. Has been receiving erlotinib, gefitinib, or afatinib for at least 6 weeks with well-controlled related toxicities less than Grade 3 in severity at the time of screening period.
6. Has radiological documentation of disease progression while receiving continuous treatment with erlotinib, gefitinib, afatinib, or osimertinib.
7. Has at least one measurable lesion per RECIST version 1.1.
8. Is willing to provide archival tumor tissue from a biopsy performed after progression during treatment with erlotinib, gefitinib, afatinib , or osimertinib OR has at least one lesion not previously irradiated, amenable to core biopsy, and is willing to undergo screening tumor biopsy.
9. Demonstrates absence of EGFR T790M. No EGFR mutation testing is required if treated with osimertinib.
10. Has Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1, with no deterioration over the previous 2 weeks.

Exclusion Criteria:

1. Has any evidence of small cell histology, or combined small cell and non-small cell histology, in original tumor biopsy or in screening biopsy performed since progression.
2. Has previously documented evidence of anaplastic lymphoma kinase (ALK) fusion, ROS proto-oncogene 1 (ROS1) fusion, BRAF V600E mutation, rearranged during transfection (RET) rearrangement, human epidermal growth factor receptor 2 (HER2) mutation, or MET exon 14 skipping mutation. No new testing for these genomic alterations is required for Screening.
3. Has received treatment with any of the following:

   1. Any cytotoxic chemotherapy, immune checkpoint inhibitor therapy, investigational agent or other anticancer drug(s) from a previous cancer treatment regimen or clinical study (other than EGFR TKI), within 14 days of the first dose of study treatment.
   2. Immune checkpoint inhibitor therapy within 30 days of first dose of study treatment.
   3. Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment.
   4. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks, or palliative radiation therapy within 2 weeks of the first dose of study drug treatment.
4. Has history of other active malignancy within 3 years prior to enrollment, except:

   1. Adequately treated non-melanoma skin cancer OR
   2. Superficial bladder tumors (tumor stage "a" [Ta], tumor stage "is" [Tis], tumor stage "1" [T1]) OR
   3. Curatively treated in situ disease OR
   4. Low risk non-metastatic prostate cancer (with Gleason score < 7, and following local treatment or undergoing active surveillance)
5. Has spinal cord compression or clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment (1 week for stereotactic radiotherapy).
6. Presence of retinal disease in the eye that is not due to neovascular age-related macular degeneration (nAMD; eg, significant diabetic retinopathy, glaucomatous retinal atrophy, retinal detachment).
7. Has history of myocardial infarction within the past 6 months.
8. Has symptomatic congestive heart failure (New York Heart Association [NYHA] Classes II-IV), unstable angina, or cardiac arrhythmia requiring antiarrhythmic treatment.
9. Has left ventricular ejection fraction (LVEF) <45% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
10. Has any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, eg, complete left bundle branch block, third-degree heart block, second-degree heart block, or PR interval >250 milliseconds (ms).
11. Has a mean QT interval corrected using Fridericia's correction (QTcF) prolongation >470 ms for females and >450 ms for males in three successive Screening measurements.
12. Unable or unwilling to discontinue concomitant use of drugs that are known to prolong the QT interval.
13. Has any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives.
14. Has any history of interstitial lung disease (pulmonary fibrosis or severe radiation pneumonitis) or is suspected to have such disease by imaging during screening.
15. Has history of pancreatitis within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (7):
- Taiwan (7):
  - Taipei Medical University, Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Jackman D, Pao W, Riely GJ, Engelman JA, Kris MG, Janne PA, Lynch T, Johnson BE, Miller VA. Clinical definition of acquired resistance to epidermal growth factor receptor tyrosine kinase inhibitors in non-small-cell lung cancer. J Clin Oncol. 2010 Jan 10;28(2):357-60. doi: 10.1200/JCO.2009.24.7049. Epub 2009 Nov 30. PMID 19949011
- [Derived] Yang JC, Su WC, Chiu CH, Shiah HS, Lee KY, Hsia TC, Uno M, Crawford N, Terakawa H, Chen WC, Takayama G, Hsu C, Hong Y, Saintilien C, McGill J, Chang GC. Evaluation of combination treatment with DS-1205c, an AXL kinase inhibitor, and osimertinib in metastatic or unresectable EGFR-mutant non-small cell lung cancer: results from a multicenter, open-label phase 1 study. Invest New Drugs. 2023 Apr;41(2):306-316. doi: 10.1007/s10637-023-01341-y. Epub 2023 Mar 9. PMID 36892745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants who met all inclusion criteria and no exclusion criteria were enrolled from 10 April 2019 to 04 September 2020 in the study at 7 clinical sites in Taiwan.
Pre-assignment Details: In the dose escalation phase, the recommended dose for expansion of DS-1205c in combination with a fixed dose of osimertinib was assessed. The doses of DS-1205c selected for this study were based on nonclinical data and were expressed in doses of DS-1205a (free base).
Groups:
- DS-1205c 200 mg + Osimertinib: Participants who received DS-1205c 200 mg twice daily (BID) at Cycle 0 monotherapy of a 7-day cycle and DS-1205c 200 mg BID in combination with 80 mg oral dose of osimertinib daily (QD) at Cycle 1 and beyond of a 21-day cycle.
- DS-1205c 400 mg + Osimertinib: Participants who received DS-1205c 400 mg twice daily (BID) at Cycle 0 monotherapy of a 7-day cycle and DS-1205c 400 mg BID in combination with 80 mg oral dose of osimertinib daily (QD) at Cycle 1 and beyond of a 21-day cycle.
- DS-1205c 800 mg + Osimertinib: Participants who received DS-1205c 800 mg twice daily (BID) at Cycle 0 monotherapy of a 7-day cycle and DS-1205c 800 mg BID in combination with 80 mg oral dose of osimertinib daily (QD) at Cycle 1 and beyond of a 21-day cycle.
- DS-1205c 1200 mg + Osimertinib: Participants who received DS-1205c 1200 mg twice daily (BID) at Cycle 0 monotherapy of a 7-day cycle and DS-1205c 1200 mg BID in combination with 80 mg oral dose of osimertinib daily (QD) at Cycle 1 and beyond of a 21-day cycle.
Period: Overall Study
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Started | 6 | 3 | 3 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 3 | 1
Not completed — Clinical progression | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Progressive disease by RECIST version 1.1 | 4 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib | Total
Number analyzed (Participants) | 6 | 3 | 3 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 2 | 0 | 7
  >=65 years | 2 | 2 | 1 | 1 | 6
Age, Continuous [Median (Full Range); unit: years] | 57.5 [45 to 77] | 73.0 [61 to 88] | 64.0 [63 to 68] | 70 [70 to 70] | 64.0 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 1 | 1 | 10
  Male | 0 | 1 | 2 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 3 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 6 | 3 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) Following Administration With DS-1205c in Combination With Osimertinib
Description: A dose-limiting toxicity (DLT) was defined as any TEAE not attributable to disease or disease-related processes that occurred during the DLT-evaluation period (Cycle 0, Day 1 to Cycle 1, Day 21 of Dose Escalation) and was Grade 3 or above, according to NCI-CTCAE Version 5.0.
Time Frame: Cycle 0, Day 1 (7-day cycle) to Cycle 1, Day 21 of Dose Escalation (each cycle was 21 days)
Population: Dose-limiting toxicities were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
Participants | 1 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Occurring in More Than 1 Participant Following Administration With DS-1205c in Combination With Osimertinib
Description: Treatment-emergent adverse events were defined as an adverse event (AE) that occurs, having been absent before the first dose of study drug, or has worsened in severity after the initiating the study drug until 30 days after last dose of the study drug.
Time Frame: Screening; Cycle 0 (7-day cycle), Days -1, 1, 2, 4, 6, and 7; Cycle 1 (21-day cycle), Days 4, 8, and 15; Cycle 2 (21-day cycle), Days 1, 2, and 8; Cycle 3 and beyond (21-day cycles), Day 1; and end-of-treatment, 30 days after last dose, up to 1 year
Population: Treatment-emergent adverse events (TEAEs) were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
Participants
  Any TEAEs | 6 | 3 | 3 | 1
  Upper respiratory tract infection | 2 | 0 | 1 | 0
  Urinary tract infection | 2 | 1 | 0 | 0
  Pneumonia | 1 | 0 | 0 | 1
  Anaemia | 0 | 1 | 1 | 1
  Insomnia | 1 | 2 | 1 | 0
  Dizziness | 1 | 1 | 0 | 0
  Headache | 1 | 0 | 1 | 0
  Cough | 1 | 1 | 0 | 0
  Dyspnoea | 1 | 1 | 0 | 0
  Haemoptysis | 1 | 1 | 0 | 0
  Vomiting | 3 | 1 | 0 | 0
  Diarrhoea | 0 | 1 | 2 | 0
  Constipation | 2 | 0 | 0 | 0
  Rash | 1 | 1 | 0 | 0
  Fatigue | 1 | 2 | 0 | 0
  Pyrexia | 0 | 0 | 2 | 0
  Alanine aminotransferase increased | 1 | 0 | 1 | 1
  Aspartate aminotransferase increased | 1 | 0 | 1 | 1
  Blood Creatinine Phosphokinase Increased | 0 | 1 | 1 | 1
  Blood Creatinine Increased | 0 | 1 | 1 | 0
  Ejection Fraction Decreased | 0 | 1 | 1 | 0
  Lipase Increased | 0 | 0 | 1 | 1
  Overdose | 0 | 0 | 2 | 0

3. Secondary Outcome: Number of Participants With Best Overall Response Assessed by Investigator Following Administration of DS-1205c in Combination With Osimertinib
Description: Complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions. Objective response rate is calculated as the number of participants with best objective response [complete response (CR) or partial response (PR) determined by Investigator assessment based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1], divided by the number of participants in the analysis population.
Time Frame: Screening; Cycle 0 (7-day cycle); Cycle 1 and beyond (21-day cycles), Every 6 weeks (± 7 days) in the first 24 weeks after Day 1 of Cycle 1, and every 12 weeks (± 7 days) thereafter; and end-of-treatment, 30 days after last dose, up to 1 year
Population: Best overall response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
Participants
  Complete response (CR) | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 0 | 0 | 0
  Stable disease (SD) | 2 | 3 | 3 | 1
  Progressive disease (PD) | 3 | 0 | 0 | 0
  Not evaluable (NE) | 1 | 0 | 0 | 0
  Overall response rate (ORR) | 0 | 0 | 0 | 0

4. Secondary Outcome: Disease Control Rate Assessed by Investigator Following Administration of DS-1205c in Combination With Osimertinib
Description: Disease control rate (DCR) is defined as the sum of complete response (CR) rate, partial response (PR) rate, and stable disease (SD) rate. As per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), complete response (CR) was defined as a disappearance of all target lesions, partial response (PR) was defined as at least a 30% decrease in the sum of diameters of target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: as for outcome 3
Population: Disease control rate was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
Participants | 2 | 3 | 3 | 1

5. Secondary Outcome: Progression-free Survival Assessed by Investigator Following Administration of DS-1205c in Combination With Osimertinib
Description: Progression-free survival is defined as the time from the date of first dose to the earliest date of the first objective documentation of disease progression or death due to any cause. As per the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 3
Population: Progression-free survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
weeks | 7.1 [5.4 to 36.6] | NA [12.3 to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. The estimated upper bound of 95% confidence interval is essentially infinity, therefore it is also N/A. | 22.0 [12.1 to 22.0] | 12.4 [NA to NA] — Not enough sample size to estimate a standard error for the median survival time so the 95% confidence interval bounds are N/A.

6. Secondary Outcome: Overall Survival in Participants Following Administration of DS-1205c in Combination With Osimertinib
Description: Overall survival was defined as the time from the date of first dose to the date of death due to any cause.
Time Frame: as for outcome 3
Population: Overall survival was assessed in the Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
weeks | 46.9 [34.0 to NA] — The estimated upper bound of 95% confidence interval is essentially infinity, therefore it is N/A. | NA [14 to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. The estimated upper bound of 95% confidence interval is essentially infinity, therefore it is also N/A. | NA [32 to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. The estimated upper bound of 95% confidence interval is essentially infinity, therefore it is also N/A. | NA [NA to NA] — Not enough sample size to estimate a standard error for the median survival time so the median and 95% confidence interval bounds are both N/A.

7. Secondary Outcome: Maximum Concentration (Cmax) Following Administration of DS-1205c Alone and in Combination With Osimertinib
Description: The maximum concentration (Cmax) of DS-1205c alone and in combination with osimertinib was assessed. Pharmacokinetic (PK) parameters for each participant were estimated using non-compartmental analysis. Descriptive statistics are provided for all plasma concentration data by analyte/dose/study day/time and for each PK parameter by analyte/dose/study day, as appropriate.
Time Frame: Predose, 1, 2, 4, 6, 8, and 12 hours of Cycle 0 (7-day cycle; DS-1205c alone), Day 1; Predose, 1, 2, 4, 6, 8, and 10 hours of Cycle 0, Day 7 (DS-1205c alone); Predose, 1, 2, 4, 6, 8, 10, and 12 hours of Cycle 2 (21-day cycle), Day 1 (DS-1205c+osimertinib)
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
ng/mL
  Cycle 0: Day 1 | 292 (94.8) | 413 (94.0) | 499 (222) | 703 (NA) — Due to small sample size, standard deviation could not be calculated.
  Cycle 0: Day 7 | 561 (191) | 827 (299) | 1041 (460) | 1070 (NA) — Due to small sample size, standard deviation could not be calculated.
  Cycle 2: Day 1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Cycle 2: Day 1 | 544 (176) | 845 (328) | 921 (260) | 1150 (NA) — Due to small sample size, standard deviation could not be calculated.

8. Secondary Outcome: Area Under the Plasma Concentration Curve Following Administration of DS-1205c Alone and in Combination With Osimertinib
Description: The area under the plasma concentration curve from time 0 until last quantifiable time point (AUClast) and the area under the plasma concentration curve over a dosing interval (AUCtau) of DS-1205c alone and in combination with osimertinib were assessed. Pharmacokinetic (PK) parameters for each participant were estimated using non-compartmental analysis. Descriptive statistics are provided for all plasma concentration data by analyte/dose/study day/time and for each PK parameter by analyte/dose/study day, as appropriate.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
h*ng/mL
  AUClast, Cycle 0: Day 1 | 1916 (530) | 2493 (277) | 2891 (1398) | 5050 (NA) — Due to small sample size, standard deviation could not be calculated.
  AUClast, Cycle 0: Day 7 | 4193 (1514) | 5716 (1931) | 7385 (4562) | 8602 (NA) — Due to small sample size, standard deviation could not be calculated.
  AUClast, Cycle 2: Day 1: number analyzed (Participants) | 5 | 3 | 3 | 1
  AUClast, Cycle 2: Day 1 | 4445 (1389) | 6852 (2716) | 7220 (2629) | 9495 (NA) — Due to small sample size, standard deviation could not be calculated.
  AUCtau, Cycle 0: Day 1 | 1975 (563) | 2557 (257) | 3002 (1472) | 5255 (NA) — Due to small sample size, standard deviation could not be calculated.
  AUCtau, Cycle 0: Day 7: number analyzed (Participants) | 6 | 3 | 1 | 1
  AUCtau, Cycle 0: Day 7 | 4818 (1772) | 6496 (2208) | 6972 (NA) — Due to small sample size, standard deviation could not be calculated. | 10300 (NA) — Due to small sample size, standard deviation could not be calculated.
  AUCtau, Cycle 2: Day 1: number analyzed (Participants) | 5 | 3 | 3 | 1
  AUCtau, Cycle 2: Day 1 | 4596 (1488) | 7117 (2883) | 7640 (2918) | 10000 (NA) — Due to small sample size, standard deviation could not be calculated.

9. Secondary Outcome: Time to Maximum Concentration (Tmax) Following Administration of DS-1205c Alone and in Combination With Osimertinib
Description: The time to maximum concentration (Tmax) of DS-1205c alone and in combination with osimertinib was assessed. Pharmacokinetic (PK) parameters for each participant were estimated using non-compartmental analysis. Descriptive statistics are provided for all plasma concentration data by analyte/dose/study day/time and for each PK parameter by analyte/dose/study day, as appropriate.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
hours
  Cycle 0: Day 1 | 4.1 [2.0 to 6.0] | 4.0 [3.9 to 4.0] | 3.9 [2.0 to 4.0] | 6.2 [6.2 to 6.2]
  Cycle 0: Day 7 | 4.0 [2.0 to 4.2] | 4.0 [2.1 to 4.0] | 4.0 [3.9 to 5.9] | 4.0 [4.0 to 4.0]
  Cycle 2: Day 1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Cycle 2: Day 1 | 4.1 [4.0 to 4.2] | 4.0 [2.0 to 4.1] | 2.1 [0 to 4.0] | 3.9 [3.9 to 3.9]

10. Secondary Outcome: Trough Plasma Concentration (Ctrough) Following Administration of DS-1205c Alone and in Combination With Osimertinib
Description: The trough plasma concentration (Ctrough) of DS-1205c alone and in combination with osimertinib was assessed. Pharmacokinetic (PK) parameters for each participant were estimated using non-compartmental analysis. Descriptive statistics are provided for all plasma concentration data by analyte/dose/study day/time and for each PK parameter by analyte/dose/study day, as appropriate.
Time Frame: as for outcome 7
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 6 | 3 | 3 | 1
ng/mL
  Cycle 0: Day 7 | 376 (143) | 460 (219) | 688 (631) | 816 (NA) — Due to small sample size, standard deviation could not be calculated.
  Cycle 2: Day 1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Cycle 2: Day 1 | 359 (137) | 576 (275) | 722 (406) | 903 (NA) — Due to small sample size, standard deviation could not be calculated.

11. Secondary Outcome: Terminal Half-life (t1/2) Following Administration of DS-1205c Alone and in Combination With Osimertinib
Description: The terminal half-life (t1/2) of DS-1205c alone and in combination with osimertinib was assessed. Pharmacokinetic (PK) parameters for each participant were estimated using non-compartmental analysis. Descriptive statistics are provided for all plasma concentration data by analyte/dose/study day/time and for each PK parameter by analyte/dose/study day, as appropriate.
Time Frame: as for outcome 7
Population: The pharmacokinetic parameter of terminal half-life (t1/2) was assessed in the Pharmacokinetic Analysis Set, except for 1 patient (Cohort 1) who did not have an available sample.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
Number analyzed (Participants) | 5 | 3 | 3 | 1
hours
  Cycle 0: Day 1 | 6.98 (1.89) | 5.3 (1.0) | 4.7 (0.6) | 3.3 (NA) — Due to small sample size, standard deviation could not be calculated.
  Cycle 0: Day 7: number analyzed (Participants) | 4 | 2 | 1 | 0
  Cycle 0: Day 7 | 11.6 (6.7) | 7.1 (1.0) | 6.9 (NA) — Due to small sample size, standard deviation could not be calculated. |
  Cycle 2: Day 1: number analyzed (Participants) | 3 | 3 | 3 | 1
  Cycle 2: Day 1 | 9.8 (3.3) | 7.9 (0.8) | 7.0 (1.3) | 11.7 (NA) — Due to small sample size, standard deviation could not be calculated.

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected at Screening, Cycle 0 (7-day cycle), Days -1, 1, 2, 4, 6, and 7; Cycle 1 (21-day cycle), Days 4, 8, and 15; Cycle 2 (21-day cycle), Days 1, 2, and 8; Cycle 3 and beyond (21-day cycles), Day 1; and end-of-treatment, 30 days after last dose, up to 1 year.
Description: A TEAE is defined as an adverse event that occurs, having been absent before the first dose of study drug, or has worsened in severity after the initiation of the study drug until 30 days after last dose of the study drug.
Arm/Group | DS-1205c 200 mg + Osimertinib | DS-1205c 400 mg + Osimertinib | DS-1205c 800 mg + Osimertinib | DS-1205c 1200 mg + Osimertinib
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/3 | 2/3 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1205c 200 mg + Osimertinib (N=6) | DS-1205c 400 mg + Osimertinib (N=3) | DS-1205c 800 mg + Osimertinib (N=3) | DS-1205c 1200 mg + Osimertinib (N=1)
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-1205c 200 mg + Osimertinib (N=6) | DS-1205c 400 mg + Osimertinib (N=3) | DS-1205c 800 mg + Osimertinib (N=3) | DS-1205c 1200 mg + Osimertinib (N=1)
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 1 | 1 | 0
Haemopytsis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Breath sounds abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cornea verticillata (Eye disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematuria (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated based on a business decision by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03255083/Prot_SAP_000.pdf